CLINICAL TRIAL: NCT07288632
Title: Effects of Genomic Profiles on Thromboembolic Risk in Patients With Locally Advanced or Metastatic Non-small-cell Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: University Of Perugia (Other)
Responsible Party: Principal Investigator, MELINA VERSO, Associate Professor, University Of Perugia
Other Study IDs: 20223ZYAJL
Record Dates: First submitted 2025-09-04; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-09

CONDITIONS: Venous Thromboembolism (VTE); NSCLC (Advanced Non-small Cell Lung Cancer)
Keywords: NSCLC; venous thromboembolism; genomic profile; activation of coagulation cascade
MeSH Terms: conditions — Venous Thromboembolism; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — levels of plasma TF, thrombin generation, IL 6, vWF, ADAMTS-13 activity PAI-1 and soluble P-selectin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with diagnosis of locally advanced or metastatic NSCLC: NSCLC patients will be enrolled in the study with a ratio 1:1 for oncogene addicted or wild type group. The oncogene-addicted group (Group A): patients with at least one oncogene mutation (ie. patients expressing EGFR mutations, KRAS mutation, ALK or ROS1 rearrangements); the wild type group (Group B): patients without oncogene mutations, categorized in 2 subgroups according to expression of PD1/PD-L1 mutation or not.

SUMMARY:
Multicenter, prospective observational study (15 Oncologic Centers, in Italy). The purpose of the study is to assess the thromboembolic potential in patients with oncogene-addicted and wild-type NSCLC. The primary aim of this project is to evaluate the association between oncogene mutations and levels of plasma parameters of the activated coagulation cascade as the plasma levels of TF, thrombin generation, IL 6, vWF, ADAMTS-13 activity, PAI-1, and soluble P-selectin in NSCLC patients. A total of 500 NSCLC patients with a diagnosis (cytologically or histologically confirmed) of locally advanced or metastatic disease will be enrolled in the study, with a ratio of 1:1 for oncogene addicted or wild-type group. The oncogene-addicted group (Group A): patients with at least one oncogene mutation (i.e., patients expressing EGFR mutations, KRAS mutation, ALK or ROS1 rearrangements); the wild type group (Group B): patients without oncogene mutations, categorized in 2 subgroups according to expression of PD1/PD-L1 mutation or not. Patients will be followed up prospectively for 6 months or until death, VTE event, loss to follow-up, or voluntary consent withdrawal.

This study will evaluate the effects of EGFR, KRAS mutations and ALK/ROS 1 and PD-1/PD-L1 rearrangements on the expression of TF and thrombin generation or the interaction between inflammation and endothelial or platelet and cancer cells, in patients with NSCLC. The study will also evaluate the potential correlation between VTE events and the expression of oncogene mutations in patients with NSCLC.

The results of this study could generate the hypothesis of including the genetic profile as variable for a risk-stratification tools and decision-making algorithms in NSCLC patients.

DETAILED DESCRIPTION:
The primary outcome is to determine the levels of plasma TF, thrombin generation, IL6, vWF, ADAMTS-13 activity, PAI-1, and soluble P-selectin in patients with NSCLC before starting the new line of anticancer therapy and after 3 and 6 months of anticancer treatment, across different patterns and association of oncogene mutations.

The further endpoints of the study will be to evaluate:

* Levels of plasma TF, thrombin generation, IL6, vWF, ADAMTS-13 activity, PAI-1, and soluble P-selectin across different cancer stages and oncogene profile;
* The potential correlation between VTE events with Levels of plasma TF, thrombin generation, IL6, vWF, ADAMTS-13 activity, PAI-1, and soluble P-selectin;
* VTE risk across different patterns of oncogene mutations in NSCLC patients;
* Role of combined strategies including clinical patients' features, Levels of plasma TF, thrombin generation, IL6, vWF, ADAMTS-13 activity, PAI-1, and soluble P-selectin and oncogene mutations to assess the risk of VTE in patients with NSCLC;
* Role of anticancer treatments in modifying the rate of clinically overt VTE events in patients with oncogene addicted or wild-type pattern of NSCLC,
* Analysis of survival based on oncogenic profile and Levels of plasma TF, thrombin generation, IL6, vWF, ADAMTS-13 activity, PAI-1, and soluble P-selectin.

Blood sampling:

Levels of plasma TF, thrombin generation, IL6, vWF, ADAMTS-13 activity, PAI-1, and soluble P-selectin in patients with NSCLC before starting the anticancer therapy, at 3 months, and at 6 months, or in case of clinical suspicion of symptomatic VTE event, or documented incidental proximal deep vein thrombosis, or pulmonary embolism will be collected.

Each collected blood sample will be collected and stocked at each participating center, and subsequently all collected blood samples will be sent for laboratory analysis.

Criteria for diagnosis of VTE:

During follow-up visits, occurrence, and clinical features of objectively confirmed VTE events will be recorded, such as the presence of symptoms and sign of proximal deep vein thrombosis (DVT) or pulmonary embolism (PE), location of VTE. The time from the diagnosis of lung cancer and the occurrence of VTE will also be recorded.

VTE event will be defined as an objectively confirmed VTE episode, which includes proximal deep-vein thrombosis of the lower limbs (symptomatic or incidental), symptomatic deep-vein thrombosis of the upper limbs, and pulmonary embolism (symptomatic, incidental, or fatal) occurring during the 6 months follow-up period.

The criteria for proximal DVT diagnosis will be the presence of a new filling defect in the iliac, femoral, or popliteal veins, in the vena cava veins, or in the axillary, or subclavian veins.

The criteria for PE diagnosis will be the presence of a new filling defect in the pulmonary arteries that will be classified as central, lobar, segmental, or sub-segmental, according to the location of emboli.

Incidental DVT or PE will be thromboembolic events detected on imaging tests performed for reasons other than clinical suspicion of VTE (i.e., imaging performed for cancer re-staging). Incidental PE will be considered with a filling defect involving a segmental or more proximal pulmonary artery.

An independent adjudication committee of vascular and radiological experts, with the scope to confirm or rule out diagnosis and classify the cause of the deaths as VTE-related or not VTE-related.

Duration of enrollment: 36 months Follow-up: Patients will be followed up prospectively for 6 months or until death, VTE event, loss to follow-up, or voluntary consent withdrawal.

Visits at enrollment and 3 and 6 months will be scheduled. Additional visits will be provided in case of clinical suspicion of symptomatic VTE event or in case of documented incidental proximal lower limb deep vein thrombosis or pulmonary embolism.

Data analysis: Characteristics of patients were described by mean, SD, median, first and third quartiles for continuous variables and by frequencies and percentages for categorical variables.

Differences in patient characteristics between the two groups will be analyzed with descriptive statistics. The study outcomes will be reported according to pre-categorized groups. The association between specific oncogene mutations and the occurrence of VTE events will also be analyzed.

A competing risk analysis will be performed to determine the cumulative incidence of VTE with death considered a competing event. Cumulative incidences will be presented as a proportion with a 95% confidence interval. Gray's test will be used to identify statistically significant differences between different groups. Overall survival rate will be analyzed by the Kaplan-Meier survival curve, and the differences among groups were assessed by the log-rank test.

Time-to-outcome event will be analyzed using a Cox proportional hazards model that includes predefined groups.

An event-free survival analysis will also be performed. Event-free survival will be defined as the absence of VTE and death.

All statistical tests will be two-sided and P value <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* • Patients aged 18 years or older,

  * Cytological or histological confirmation of NSCLC,
  * Locally advanced or metastatic disease (Stage III-IV),
  * Patients starting a new anticancer treatment for locally advanced/metastatic disease (first or further line of treatment),
  * Testing for oncogenic (EGFR, KRAS, ALK, ROS1 and PD-1/PD-L1) profile performed,
  * Written informed consent

Exclusion Criteria:

* • Patients received surgery or radiotherapy for lung cancer within the past 3 months before recruitment or chemotherapy within the past 1 months before recruitment,

  * Patients with a history of VTE after cancer diagnosis or evidence of VTE events at enrollment
  * Continuative use of anticoagulant drugs for any indication (atrial fibrillation or previous VTE)
  * ECOG performance profile 3 or 4
  * Life expectancy of less than 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis (cytologically or histologically confirmed) of locally advanced or metastatic disease will be enrolled in the study with a ratio 1:1 for oncogene addicted or wild type group.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-02-09 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Levels of plasma TF, thrombin generation, IL6, vWF, ADAMTS-13 activity, PAI-1and soluble P-selectin | From enrollment to the end of study period at 6 months
  Levels of plasma TF, thrombin generation, IL6, vWF, ADAMTS-13 activity, PAI-1and soluble P-selectin in patients with NSCLC before the starting of the new line of anticancer therapy and after 3 and 6 months of anticancer treatment, across different patterns and association of oncogene mutations.

CONTACTS AND LOCATIONS:
Overall Officials: Melina Verso, Principal Investigator — Univesity of Perugia
Locations (1):
- Emily Oliovecchio, Perugia, Perugia, Italy

IPD SHARING:
Plan to Share IPD: No
IPD will be share only with the co-Investigators

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-05-30): https://cdn.clinicaltrials.gov/large-docs/32/NCT07288632/Prot_SAP_000.pdf
  • Informed Consent Form (2025-05-30): https://cdn.clinicaltrials.gov/large-docs/32/NCT07288632/ICF_001.pdf